CLINICAL TRIAL: NCT05441683
Title: Comparison of Vertical Releasing Incisions and Horizontal Extending Incisions for Periodontal Accelerated Osteogenic Orthodontics in the Anterior Region: A Randomized Controlled Trial With Surgical Time, Clinical and Radiographic Outcomes
Brief Title: Comparing of the Clinical Outcome of Periodontal Accelerated Osteogenic Orthodontics With Horizontal or Vertical Releasing Incisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0271
Record Dates: First submitted 2022-06-13; First posted 2022-07-01 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Malocclusion
Keywords: periodontal accelerated osteogenic orthodontics; vertical releasing incision
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEI group (Experimental): PAOO with horizontal extending incisions on both sides
  Interventions: Procedure: horizontal extending incision
- VRI group (Active Comparator): PAOO with vertical releasing incisions on both sides
  Interventions: Procedure: vertical releasing incision

INTERVENTIONS:
Procedure: horizontal extending incision — a papilla preserving incision will be made on the labial side of the front teeth with a thin alveolar bone or dehiscence and/or fenestration. Then horizontally extending incisions will be added to each side of the initial incision, extending one to two teeth beyond the defected area, before a full-thickness flap is lifted.
  Arms: HEI group
Procedure: vertical releasing incision — a papilla preserving incision will be made on the labial side of the front teeth with a thin alveolar bone or dehiscence and/or fenestration. Vertical releasing incisions will be made on each side of the initial incision before a full-thickness flap is lifted. The incision formed an oblique trapezoidal flap with a wider base.
  Arms: VRI group

SUMMARY:
The study aims to compare the effect of periodontal accelerated osteogenic orthodontics (PAOO) with horizontal or vertical releasing incisions on operation time, healing, adverse effects, and effectiveness of bone augmentation.

Methods: A total of 22 patients requiring PAOO surgery due to orthodontic treatment were enrolled in this trial, and randomly divided into test or control group, consisting of 11 subjects in each. The test group will receive PAOO with horizontal extending incisions on both sides of the flap; while the control group will receive PAOO with vertical releasing incisions; the two groups use the same surgical technic except for the incision design. Outcome measures include: operation time, postoperative scar, radiographic data (alveolar height and alveolar ridge thickness), gingival thickness, etc. Clinical evaluation will be performed at 1 week, 2 weeks, 3months, 6 months and 12 months after operation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 40 years old, systemic healthy, undergoing or planning to undergo orthodontic treatment.
2. Patients with a thin alveolar bone or with dehiscence and/or fenestration on the labial side of maxillary or mandibular front teeth area.
3. Patients with expected tooth movement beyond the labial alveolar bone during orthodontic procedures.

Exclusion Criteria:

1. Smoker.
2. Pregnant or lactating.
3. Untreated periodontitis.
4. Presence of <2mm keratinized gingival width(KGW) or thin gingival phenotype (as defined by dental probe transparency.)
5. History of orthodontic and/or orthognathic treatment.
6. With systemic disease (diabetes, hypertension, heart disease, malignant tumor, severe mental illness, and other surgical contraindications.)
7. Long-term medication (immunosuppressive drugs, bisphosphonates, etc.)
8. Poor adherence to complete one-year follow-up.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanmin Wu, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: teeth
Groups:
- HEI Group: PAOO with horizontally extending incisions on both sides
  horizontally extending incisions (HEIs): a papilla preserving incision will be made on the labial side of the front teeth with a thin alveolar bone or dehiscence and/or fenestration. Then horizontally extending incisions will be added to each side of the initial incision, extending one to two teeth beyond the defected area, before a full-thickness flap is lifted.
- VRI Group: PAOO with vertical releasing incisions on both sides
  Vertical releasing incisions (VRIs):a papilla preserving incision will be made on the labial side of the front teeth with a thin alveolar bone or dehiscence and/or fenestration. Vertical releasing incisions will be made on each side of the initial incision before a full-thickness flap is lifted. The incision formed an oblique trapezoidal flap with a wider base.
Period: Overall Study
Arm/Group | HEI Group | VRI Group
Started | 11; 66 teeth | 11; 63 teeth
Completed | 10; 60 teeth | 10; 57 teeth
Not Completed | 1; 6 teeth | 1; 6 teeth

BASELINE CHARACTERISTICS:
Population: A total of 22 participants were enrolled between July 2022 and August 2023. Following randomization, one participant in the VRI group was excluded due to postoperative smoking, and one in the HEI group dropped out because of a second surgery. Each participant could contribute up to six anterior teeth as analysis units. In total, 20 patients and 117 anterior teeth were included. Two central incisors and one lateral incisor were congenitally missing in two participants.
Units Other Than Participants: teeth
Groups:
- HEI Group: Periodontal Accelerated Osteogenic Orthodontics (PAOO) with horizontally extending incisions on both sides
  horizontally extending incision: a papilla preserving incision will be made on the labial side of the front teeth with a thin alveolar bone or dehiscence and/or fenestration. Then horizontally extending incisions will be added to each side of the initial incision, extending one to two teeth beyond the defected area, before a full-thickness flap is lifted.
- VRI Group: Periodontal Accelerated Osteogenic Orthodontics (PAOO) with vertical releasing incisions on both sides
  vertical releasing incision: a papilla preserving incision will be made on the labial side of the front teeth with a thin alveolar bone or dehiscence and/or fenestration. Vertical releasing incisions will be made on each side of the initial incision before a full-thickness flap is lifted.
- Total: Total of all reporting groups
Arm/Group | HEI Group | VRI Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Number analyzed (teeth) | 60 | 57 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.20 (4.64) | 27.20 (5.07) | 27.20 (4.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Surgery Time
Description: Timing will start when the first incision is about to be made, and end when the last suture is complete. The time in between will be recorded as surgery time.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
minutes | 57.66 (5.01) | 68.50 (13.50)

2. Secondary Outcome: Probing Depth (PD)
Description: Distance from gingival margin to base of periodontal pocket. It will be measured at baseline and 3 months, 6 months, and 12months after surgery.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: teeth
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Number analyzed (teeth) | 60 | 57
millimeter
  baseline | 1.86 (0.32) | 1.86 (1.83)
  3 months change | -0.05 (0.45) | 0.06 (0.42)
  6 months change | 0.03 (0.43) | 0.13 (0.56)
  12 months change | -0.07 (0.58) | -0.05 (0.59)

3. Secondary Outcome: Clinical Attachment Level (CAL)
Description: Distance from CEJ to base of periodontal pocket. It will be measured at baseline and 3 months, 6 months, and 12months after surgery.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: teeth
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Number analyzed (teeth) | 60 | 57
millimeter
  baseline | 0.66 (1.05) | 0.52 (0.89)
  3 months change | 0.05 (0.77) | 0.05 (0.75)
  6 months change | 0.01 (0.80) | 0.16 (0.76)
  12 months change | 0.15 (0.85) | -0.15 (0.78)

4. Secondary Outcome: Keratinized Gingival Width (KGW)
Description: From mucogingival junction to free gingival margin It will be measured at baseline and 3 months, 6 months, and 12months after surgery.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: teeth
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Number analyzed (teeth) | 60 | 57
millimeter
  baseline | 2.97 (0.72) | 3.50 (1.30)
  3 months change | 0.50 (0.86) | 0.07 (1.39)
  6 months change | 0.37 (1.12) | 0.41 (1.38)
  12 months change | 0.85 (1.13) | 0.71 (1.15)

5. Secondary Outcome: Gingival Recession Depth (GRD)
Description: Distance from CEJ to gingival margin. It will be measured at baseline and 3 months, 6 months, and 12months after surgery.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: teeth
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Number analyzed (teeth) | 60 | 57
millimeter
  baseline | -0.75 (1.03) | -0.96 (1.25)
  3 months change | -0.06 (0.77) | 0.14 (0.67)
  6 months change | -0.08 (0.99) | 0.21 (0.70)
  12 months change | -0.04 (0.89) | 0.01 (0.77)

6. Secondary Outcome: Root Length
Description: the distance from the CEJ to the apex of the root. It will be measured at baseline, 6 months, and 12months after surgery.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: teeth
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Number analyzed (teeth) | 60 | 57
millimeter
  baseline | 11.11 (1.81) | 12.03 (2.45)
  6 months change | -0.30 (0.78) | -0.45 (1.09)
  12 months change | -0.44 (1.00) | -064 (1.09)

7. Secondary Outcome: Vertical Bone Height (VBL)
Description: the distance from the cemento-enamel junction to the crest of the labial alveolar bone.
  It will be measured at baseline, 6 months, and 12months after surgery.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: teeth
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Number analyzed (teeth) | 60 | 57
millimeter
  baseline | 4.28 (2.99) | 5.06 (3.00)
  6 months change | -2.95 (2.75) | -3.17 (2.76)
  12 months change | -2.69 (2.96) | -2.94 (2.79)

8. Secondary Outcome: Alveolar Bone Width Measured at 2 mm Below the CEJ (BW2)
Description: Alveolar bone width measured at 2 mm below the CEJ on the labial side of the alveolar bone, representing the distance from the tooth root surface to the labial bone surface.It will be measured at baseline, 6 months, and 12months after surgery.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: teeth
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Number analyzed (teeth) | 60 | 57
millimeter
  baseline | 0.33 (0.47) | 0.18 (0.40)
  6 months change | 0.80 (0.86) | 0.45 (0.69)
  12 months change | 0.67 (0.78) | 0.39 (0.67)

9. Secondary Outcome: Alveolar Bone Width Measured at 4 mm Below the CEJ (BW4)
Description: Alveolar bone width measured at 4 mm below the CEJ on the labial side of the alveolar bone, representing the distance from the tooth root surface to the labial bone surface.It will be measured at baseline, 6 months, and 12months after surgery.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: teeth
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Number analyzed (teeth) | 60 | 57
millimeter
  baseline | 0.43 (0.48) | 0.39 (0.50)
  6 months change | 1.71 (1.00) | 0.96 (0.68)
  12 months change | 1.44 (0.73) | 0.94 (0.51)

10. Secondary Outcome: Alveolar Bone Width Measured at 6 mm Below the CEJ (BW6)
Description: Alveolar bone width measured at 6 mm below the CEJ on the labial side of the alveolar bone, representing the distance from the tooth root surface to the labial bone surface.It will be measured at baseline, 6 months, and 12months after surgery.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: teeth
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Number analyzed (teeth) | 60 | 57
millimeter
  baseline | 0.45 (0.50) | 0.51 (0.46)
  6 months change | 2.47 (1.11) | 1.38 (0.85)
  12 months change | 1.92 (0.87) | 1.13 (0.68)

11. Secondary Outcome: Number of Participants With Visible Scarring
Description: Gingival scarring was evaluated at 12 months postoperatively through visual inspection. Participants were classified as scar-positive if any visible scar was present at the surgical site, including normotrophic scars (flat and white) and pathological scars (raised or irregular in shape).
  Each participant was counted once regardless of scar characteristics.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Participants | 1 | 6

12. Secondary Outcome: Pain Level
Description: measured with visual analogue score (VAS): 0 (no pain/normal sensation) to 10 (intolerable pain/complete numbness)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
score on a scale
  1 week | 2.90 (1.20) | 2.70 (1.16)
  2 weeks | 1.60 (1.08) | 1.50 (1.08)

13. Secondary Outcome: Membrane Exposure
Description: membrane exposure was observed and assessed as a binary outcome (yes/no). Recorded "no" if there is no membrane exposure, and "yes" if there is any membrane exposure.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Participants
  yes | 3 | 1
  no | 7 | 9

14. Secondary Outcome: Facial Swelling
Description: recorded "0" for no facial swelling; "1" for mild facial swelling; "2" for severe facial swelling. It will be measured at 1 and 2 weeks after surgery.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Participants
  1 week: 0 | 6 | 4
  1 week: 1 | 4 | 6
  1 week: 2 | 0 | 0
  2 weeks: 0 | 10 | 10
  2 weeks: 1 | 0 | 0
  2 weeks: 2 | 0 | 0

15. Secondary Outcome: Mucosal Color
Description: recorded "0" for no redness along the incision; "1" for slight redness; "2" for obvious redness. It will be measured at 1 and 2 weeks after surgery.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Participants
  1 week: 0 | 0 | 0
  1 week: 1 | 10 | 9
  1 week: 2 | 0 | 1
  2 weeks: 0 | 0 | 1
  2 weeks: 1 | 10 | 9
  2 weeks: 2 | 0 | 0

16. Secondary Outcome: Mucosa Edema
Description: recorded "0" for no edema around the surgery area; "1" for mild edema; "2" for severe edema.It will be measured at 1 and 2 weeks after surgery.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
Participants
  1 week: 0 | 1 | 0
  1 week: 1 | 7 | 6
  1 week: 2 | 2 | 4
  2 weeks: 0 | 3 | 3
  2 weeks: 1 | 7 | 7
  2 weeks: 2 | 0 | 0

17. Other Pre Specified Outcome: Particulate Bone Grafting Material Weight
Description: The net weight of the bone graft material before surgery is recorded as W1. After surgery, the remaining bone graft material was collected, dried, and weighed by the same electronic scale as W2. The amount of bone graft material used during surgery was calculated as ΔW=W1-W2.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: g
Arm/Group | HEI Group | VRI Group
Number analyzed (Participants) | 10 | 10
g | 0.83 (0.23) | 0.79 (0.25)

ADVERSE EVENTS:
Time Frame: From baseline (pre-intervention) until 12 months after the last treatment session.
Arm/Group | HEI Group | VRI Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT05441683/Prot_SAP_000.pdf